CLINICAL TRIAL: NCT02212899
Title: Prospective, Observational Registry of Renaissance-guided Spine Surgeries
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Mazor Robotics (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN111
Record Dates: First submitted 2014-05-11; First posted 2014-08-08 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Degenerative Spine Disease; Spinal Deformity
Keywords: Spinal Surgery; Spinal Fusion; Deformity Correction; Spinal Instrumentation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
To establish an observational registry for systematic collection of clinical data from Renaissance-guided spine surgeries.

DETAILED DESCRIPTION:
The key objective of this observational registry is to prospectively collect data to facilitate the quantification of potential short- and long-term benefits of Renaissance-guided spine surgery. It establishes a common framework for collaboration between surgeons performing Renaissance-guided spine surgeries in either minimally invasive (MIS) or open surgical approaches.

The main endpoints that will be collected are surgical endpoints (e.g. complication rates), patient reported outcomes (e.g. VAS, ODI), imaging parameters (e.g. coronal and sagittal alignment, mainly in reconstructive surgeries for spinal deformities) and technical parameters (e.g. use of intraoperative fluoroscopy, ratio of planned vs. executed screws).

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing spinal surgery in a posterior approach where the surgeon used Renaissance surgical guidance system.

Patient capable of complying with study requirements. Signed informed consent by patient.

Exclusion Criteria:

Any significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study.

Patient cannot follow study protocol, for any reason. Patient cannot or will not sign informed consent.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any pediatric, adolescent or adult patient undergoing open or MIS Renaissance-guided spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes as measured on plain radiographs | Within 10 years of surgery
  sagittal and coronal alignment in reconstructive surgeries for spinal deformities
Surgical complications | Within 10 years of surgery
  new neural deficits, implant-related durotomy, infection requiring return to surgery, excessive blood loss
Reoperation rates | Within 10 years of surgery
  Any revision surgery on the segment of interest
Radiation exposure | Day of surgery
  Reading of exposure in seconds (and KvP if available) from C-arm or other imaging system used in the operating room

SECONDARY OUTCOMES:
Clinical performance of instrumentation technique | Day of surgery
  implant instrumentation time, total surgery time
Ratio of executed vs. planned screws | Day of surgery
  Number of screws planned for Renaissance-guided insertion, but instead inserted manually, and cause
Number of abandoned screws | Day of surgery
  the number of screws not instrumented and the reason
Neuromonitoring events | Day of surgery
Length of convalescence | within 2 years of surgery
  Length of hospital stay, destination at discharge, time to return to work, time to return to normal activities
Improvement in health-related quality of life metrics | up to 10 years post-operative
  back and leg VAS, Oswestry Disability Index (ODI), SRS22, EQ-5D-5L, in accordance with the surgeon's practices
Fusion rates/pseudoarthrosis | Within 1 year of surgery
  The rate of fusion as determined within one year of surgical procedure.
Implant placement accuracy | Within one year post-surgery
  Accuracy of implants as measured on a post-operative CT scan (when available)

CONTACTS AND LOCATIONS:
Overall Officials: Doron Dinstein, MD, MBA, Study Director — Mazor Robotics
Locations (4):
- United States (4):
  - Lyerly Baptist/ Lyerly Neurosurgery, Jacksonville, Florida
  - Tabor Orthopedics, Memphis, Tennessee
  - Spine Associates, Houston, Texas
  - The Virginia Spine Institute, Reston, Virginia

REFERENCES:
- [Background] Lieberman IH, Hardenbrook MA, Wang JC, Guyer RD. Assessment of pedicle screw placement accuracy, procedure time, and radiation exposure using a miniature robotic guidance system. J Spinal Disord Tech. 2012 Jul;25(5):241-8. doi: 10.1097/BSD.0b013e318218a5ef. PMID 21602728
- [Background] Devito DP, Kaplan L, Dietl R, Pfeiffer M, Horne D, Silberstein B, Hardenbrook M, Kiriyanthan G, Barzilay Y, Bruskin A, Sackerer D, Alexandrovsky V, Stuer C, Burger R, Maeurer J, Donald GD, Schoenmayr R, Friedlander A, Knoller N, Schmieder K, Pechlivanis I, Kim IS, Meyer B, Shoham M. Clinical acceptance and accuracy assessment of spinal implants guided with SpineAssist surgical robot: retrospective study. Spine (Phila Pa 1976). 2010 Nov 15;35(24):2109-15. doi: 10.1097/BRS.0b013e3181d323ab. PMID 21079498
- [Background] Kantelhardt SR, Martinez R, Baerwinkel S, Burger R, Giese A, Rohde V. Perioperative course and accuracy of screw positioning in conventional, open robotic-guided and percutaneous robotic-guided, pedicle screw placement. Eur Spine J. 2011 Jun;20(6):860-8. doi: 10.1007/s00586-011-1729-2. Epub 2011 Mar 8. PMID 21384205
- [Background] Hu X, Ohnmeiss DD, Lieberman IH. Robotic-assisted pedicle screw placement: lessons learned from the first 102 patients. Eur Spine J. 2013 Mar;22(3):661-6. doi: 10.1007/s00586-012-2499-1. Epub 2012 Sep 14. PMID 22975723
- [Background] Kosmopoulos V, Schizas C. Pedicle screw placement accuracy: a meta-analysis. Spine (Phila Pa 1976). 2007 Feb 1;32(3):E111-20. doi: 10.1097/01.brs.0000254048.79024.8b. PMID 17268254
- [Background] Rajasekaran S, Vidyadhara S, Ramesh P, Shetty AP. Randomized clinical study to compare the accuracy of navigated and non-navigated thoracic pedicle screws in deformity correction surgeries. Spine (Phila Pa 1976). 2007 Jan 15;32(2):E56-64. doi: 10.1097/01.brs.0000252094.64857.ab. PMID 17224800
- [Background] Tian NF, Huang QS, Zhou P, Zhou Y, Wu RK, Lou Y, Xu HZ. Pedicle screw insertion accuracy with different assisted methods: a systematic review and meta-analysis of comparative studies. Eur Spine J. 2011 Jun;20(6):846-59. doi: 10.1007/s00586-010-1577-5. Epub 2010 Sep 23. PMID 20862593
- [Background] Hamilton DK, Smith JS, Sansur CA, Glassman SD, Ames CP, Berven SH, Polly DW Jr, Perra JH, Knapp DR, Boachie-Adjei O, McCarthy RE, Shaffrey CI; Scoliosis Research Society Morbidity and Mortality Committee. Rates of new neurological deficit associated with spine surgery based on 108,419 procedures: a report of the scoliosis research society morbidity and mortality committee. Spine (Phila Pa 1976). 2011 Jul 1;36(15):1218-28. doi: 10.1097/BRS.0b013e3181ec5fd9. PMID 21217448